CLINICAL TRIAL: NCT01511042
Title: Non-Modulation Phenotype and Vascular Dysfunction in Diabetes Mellitus
Brief Title: Vascular Dysfunction in Diabetes: Genes and Hormones
Status: Terminated | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gordon H. Williams, MD, Chief, Cardiovascular Endocrinology Section, Brigham and Women's Hospital
Other Study IDs: 1999P001983
Record Dates: First submitted 2011-07-19; First posted 2012-01-18 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — p-Aminohippuric Acid; Angiotensin II; Norepinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Urine, blood, DNA
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Para-aminohippuric Acid — Aminohippurate sodium is an agent to measure effective renal plasma flow (ERPF). It is the sodium salt of para-aminohippuric acid, commonly abbreviated "PAH".
  Other Names: PAH
Drug: Angiotensin II — Angiotensin II (Ang II) is a naturally occurring hormone whose primary purpose is to regulate the body's internal volume. It accomplishes this task by influencing the function of a variety of organs and tissues. It increases aldosterone secretion from the adrenal gland. It causes blood vessels to contract, particularly renal blood vessels, and it modifies the way the heart works.
  Other Names: AngII; AII
Drug: Norepinephrine — A hormone that is normally present in your body, which regulates your blood pressure.
  Other Names: NE

SUMMARY:
The investigators are very excited that the National Institutes of Health are sponsoring us to investigate why patients with diabetes are more likely to develop high blood pressure, atherosclerosis (hardening of the arteries), and heart disease. There are two parts of our research program. The first part is a screening visit. At this visit you will be given a brief physical exam and will be asked questions concerning your medical history. During the same visit you will have your blood drawn for routine screening and to prepare DNA for genetic testing. You will also be asked to collect a urine sample for routine screening.

If the doctor finds that you are a healthy candidate you will be invited to participate in the second part of the study. During Phase II the investigators will perform physiologic tests after you are placed on a low salt diet and again after you are placed on a high salt diet. All of the food that you will eat during the two diets will be provided to you by the hospital. If you are on blood pressure medication, it may be necessary to discontinue taking your present medication for up to three months before beginning the study. Patients discontinuing their current blood pressure medication may be placed on a different blood pressure medication during this washout period if necessary to maintain blood pressure at pre-study levels. The investigators will take you off all medications, except cholesterol medications two weeks prior to your scheduled in-patient study. However, if you are currently on medication to control your diabetes you will remain on this throughout the entire study.

Once your blood pressure medications are discontinued, you will be closely monitored to make sure you do not encounter any difficulty. If you do not own a home blood pressure monitor, the investigators will provide one for to use during the study so that you can keep a daily record of your blood pressure readings. The investigators will ask you to call us every three days to report your blood pressure readings. Less than 20% of patients with hypertension have any significant increase in their blood pressure during this short time off therapy. After you have been off your medication for nine days the dieticians will give you low salt meals to eat at home for six days. On the sixth day of the low salt diet, you will be asked to begin a 24-hour urine collection. You will also be required to come to the Ambulatory Clinical Center (221 Longwood Ave.) for a one-hour test. You will return that evening to the inpatient Clinical Research Center where you will be admitted for your first study that will occur the next morning. On the morning of your low salt study you will have three naturally occurring hormones administered and blood samples drawn from an intravenous needle. The investigators will also take ultrasound pictures of your heart to see how salt and hormones affect the way the heart functions. These tests will last approximately five hours and you will be discharged around 12:00 p.m. The dieticians will then give you your meals for the next week to take home. Each of these meals will have a high salt content. After six days of your high salt diet, on the morning of your second admission to the hospital, you will be asked to begin a final 24-hour urine collection. The same study that was done for the low salt study will be repeated for the high salt study. You will be discharged around 3:00 p.m. This study will determine if you are salt-sensitive. A high salt diet has been found to lead to higher blood pressure and weight gain. In addition, the investigators hope to learn more about the hormones that regulate your blood pressure and the genes responsible for regulating those hormones.

You will be placed back on your initial blood pressure medication (if you are on any) and returned to your regular physician for care. The investigators will provide clinically relevant information to you and your physician.

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetes Mellitus
* Age between 18-65 years
* BMI < 40
* In overall good health

Exclusion Criteria:

* History of coronary atherosclerotic disease, MI, CVA, or significant peripheral vascular disease
* BMI > 40
* Subjects with diastolic blood pressures greater than 100 mm Hg while on anti-hypertensive medications, or systolic blood pressures greater than 160 mm Hg while on anti-hypertensive medications will be excluded.
* Current alcohol or drug abuse
* Subjects taking other medications (except thyroid supplements, oral hyperglycemic agents and insulin) will be excluded
* Subjects who are on medications that cannot be discontinued such as anti-depressants, anti-seizure medications, etc that may interfere with salt and water handling will not be studied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Type II Diabetes Mellitus
  * Age between 18-65 years
  * BMI < 40
  * In overall good health
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 1999-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Frequency of Intermediate Phenotypes in Subjects with Diabetes Mellitus versus Hypertension | 10 Years
  The frequency of salt sensitive blood pressure

SECONDARY OUTCOMES:
Frequency of polymorphic variants in AGT gene in Hypertensives versus diabetics | 10 Years
  The frequency of polymorphisms in the angiotensinogen (AGT), ACE and ALDO synthase and ALAP genes in non-modulating hypertension subset.
Frequency of salt sensitive subtype in Diabetics versus hypertensives | 10 years
  Frequency of non-modulating phenotype and low renin phenotype in the salt sensitive subjects.subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon H Williams, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital- 221 Longwood Avenue, Boston, Massachusetts, United States